CLINICAL TRIAL: NCT01385371
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Grass (Phleum Pratense) Sublingual Tablet (SCH 697243) in Subjects Between 5 and 65 Years of Age, With a History of Grass Pollen-Induced Rhinoconjunctivitis, With or Without Asthma (Protocol No. P08067)
Brief Title: A Study of SCH 697243 in Participants With Grass Pollen Allergy Symptoms, With or Without Asthma (P08067)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08067; MK-7243-001 (Other: Merck Protocol ID)
Record Dates: First submitted 2011-04-06; First posted 2011-06-30 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis Allergic; Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCH 697243 (Experimental)
  Interventions: Biological: Grass (Phleum pratense) pollen allergen extract
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo for SCH 697243

INTERVENTIONS:
Biological: Grass (Phleum pratense) pollen allergen extract — One dissolving tablet sublingually once daily
  Other Names: SCH 697243
  Arms: SCH 697243
Biological: Placebo for SCH 697243 — One dissolving tablet sublingually once daily
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of grass sublingual tablet (SCH 697243) versus placebo in the treatment of grass pollen-induced allergic hayfever symptoms. Participants will receive either the sublingual grass tablet or a placebo tablet during the study. It is expected that those participants receiving the active sublingual grass tablet will have less hayfever symptoms and need less medications to treat hayfever symptoms during the grass pollen season.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical history of significant allergic rhinoconjunctivitis to grass (with or without asthma)
* Must have a positive skin prick test response to Phleum pratense (Timothy grass)
* Must be positive for specific immunoglobulin E (IgE) against Phleum pratense (Timothy grass)
* Must have an forced expiratory volume in 1 second (FEV1) of at least 70% of predicted value at

Screening

- Safety laboratory tests and vital signs conducted at the Screening Visit must be within normal

limits or clinically acceptable to the investigator/sponsor

Exclusion Criteria:

* Has a clinical history of symptomatic seasonal allergic rhinitis and/or asthma due to another allergen during or potentially overlapping the GPS
* Has a clinical history of significant symptomatic perennial allergic rhinitis and/or asthma due to an allergen to which the participant is regularly exposed
* Has received an immunosuppressive treatment within 3 months prior to the Screening Visit
* Has a clinical history of severe asthma
* Has a history of anaphylaxis with cardiorespiratory symptoms
* Has a history of self-injectable epinephrine use
* Has a history of chronic urticaria and angioedema
* Has a clinical history of chronic sinusitis during the 2 years prior to the Screening Visit
* Has current severe atopic dermatitis
* Is breast-feeding, pregnant, or intending to become pregnant
* Had previous treatment by immunotherapy with any grass pollen allergen for more than 1 month within the 5 years prior to the Screening Visit
* Ongoing treatment with any specific immunotherapy at the time of the Screening Visit
* Has a known history of allergy, hypersensitivity or intolerance to the ingredients of the study drug (except for Phleum pratense), rescue medications, or self-injectable epinephrine
* Has any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study. Specific examples include but are not limited to hypertension being treated with beta blockers, coronary artery disease, arrhythmia, stroke, ocular conditions requiring topical beta blockers, any condition requiring the use of beta blockers
* Has used any investigational drugs within 30 days of the Screening Visit
* Is participating in any other clinical study
* Is a family member of the investigational study staff conducting this study
* Is unable to meet medication washout requirements
* Is unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the GPS, which in the opinion of the investigator will compromise the data
* Has a clinically significant abnormal vital sign or laboratory value that would preclude participation in the study

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

REFERENCES:
- [Result] Maloney J, Bernstein DI, Nelson H, Creticos P, Hebert J, Noonan M, Skoner D, Zhou Y, Kaur A, Nolte H. Efficacy and safety of grass sublingual immunotherapy tablet, MK-7243: a large randomized controlled trial. Ann Allergy Asthma Immunol. 2014 Feb;112(2):146-153.e2. doi: 10.1016/j.anai.2013.11.018. Epub 2013 Dec 21. PMID 24468255
- [Derived] Nolte M, Barber D, Maloney J, Li Z, Kaur A, Galan A, Andersen JS, Nolte H. Timothy specific IgE levels are associated with efficacy and safety of timothy grass sublingual immunotherapy tablet. Ann Allergy Asthma Immunol. 2015 Dec;115(6):509-515.e2. doi: 10.1016/j.anai.2015.09.018. Epub 2015 Oct 21. PMID 26507709
- [Derived] Hebert J, Blaiss M, Waserman S, Kim H, Creticos P, Maloney J, Kaur A, Li Z, Nelson H, Nolte H. The efficacy and safety of the Timothy grass allergy sublingual immunotherapy tablet in Canadian adults and children. Allergy Asthma Clin Immunol. 2014 Oct 30;10(1):53. doi: 10.1186/1710-1492-10-53. eCollection 2014. PMID 25685162

RESULTS

PARTICIPANT FLOW:
Groups:
- SCH 697243: Participants receiving Grass (Phleum pratense) Pollen Allergen Extract
- Placebo: Participants receiving Placebo
Period: Overall Study
Arm/Group | SCH 697243 | Placebo
Started | 752 | 749
Completed | 603 | 652
Not Completed | 149 | 97
Not completed — Adverse Event | 54 | 19
Not completed — Lost to Follow-up | 16 | 16
Not completed — Withdrawal by Subject | 52 | 39
Not completed — Protocol Violation | 25 | 21
Not completed — Administrative | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 697243 | Placebo | Total
Number analyzed (Participants) | 752 | 749 | 1501
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (14.5) | 33.5 (14.5) | 33.2 (14.5)
Gender [Count of Participants; unit: Participants]
  Female | 381 | 333 | 714
  Male | 371 | 416 | 787

OUTCOME MEASURES:

1. Primary Outcome: Average Total Combined Rhinoconjunctivitis Daily Symptom Score (DSS) and Rhinoconjunctivitis Daily Medication Score (DMS) Over the Entire Grass Pollen Season (GPS)
Description: The total combined score was the sum of the rhinoconjunctivitis DSS and rhinoconjunctivitis DMS for the entire GPS (total score range: 0 to 54), with a lower score representing less rhinoconjunctivitis symptoms and use of medications.
  For rhinoconjunctivitis DSS, participants assessed a total of 6 rhinoconjunctivitis symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes, and watery eyes) each on a scale of 0 to 3 (0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms; score range: 0 to 18), with a lower score representing less rhinoconjunctivitis symptoms.
  For rhinoconjunctivitis DMS, participants reported their use of specific rescue medications with specific scores assigned to each medication (score range: 0 to 36), with a lower score representing less use of medications for rhinoconjunctivitis.
Time Frame: Entire GPS (expected average duration of 5 to 6 weeks)
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who received at least one dose of study drug and had at least one post-treatment observation for the analysis endpoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 629 | 672
score on a scale | 3.24 [0.00 to 24.10] | 4.22 [0.00 to 23.16]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Median Difference (Final Values) = -0.98, 95% CI [-1.2 to -0.4]

2. Secondary Outcome: Average Rhinoconjunctivitis DSS Over the Entire GPS
Description: For rhinoconjunctivitis DSS, participants assessed a total of 6 rhinoconjunctivitis symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes, and watery eyes) each on a scale of 0 to 3 (0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms; score range: 0 to 18), with a lower score representing less rhinoconjunctivitis symptoms.
Time Frame: Entire GPS (expected average duration of 5 to 6 weeks)
Population: The FAS population consisted of all randomized participants who received at least one dose of study drug and had at least one post-treatment observation for the analysis endpoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 629 | 672
score on a scale | 2.49 [0.00 to 18.00] | 3.13 [0.00 to 17.67]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon Rank Sum Test; Median Difference (Final Values) = -0.64, 95% CI 2-sided [-0.7 to -0.2]

3. Secondary Outcome: Average Total Combined Rhinoconjunctivitis DSS and Rhinoconjunctivitis DMS Over the Peak GPS
Description: as for outcome 1
Time Frame: Peak GPS (expected average duration of 2 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 620 | 663
score on a scale | 3.33 [0.00 to 30.88] | 4.67 [0.00 to 34.21]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Median Difference (Final Values) = -1.33, 95% CI 2-sided [-1.4 to -0.5]

4. Secondary Outcome: Average Rhinoconjunctivitis Quality of Life Questionnaire With Standardized Activities for Participants ≥12 Years of Age (RQLQ12+) Over the Peak GPS
Description: The RQLQ12+ consists of 7 domains: Activities, Sleep, Non-Nose/Eye Symptoms, Practical Problems, Nasal Symptoms, Eye Symptoms, Emotional. Participants reflect on their experience over the previous 7 days and assess 28 items on a scale of 0 to 6 (0=Not troubled, 6=Extremely troubled; score range: 0-6 [mean of all domain scores]), with a higher score indicating more significant impairment due to seasonal allergic rhinoconjunctivitis.
Time Frame: Peak GPS (expected average duration of 2 weeks)
Population: The FAS population consisted of all randomized participants ≥12 years of age who received at least one dose of study drug and had at least one post-treatment observation for the analysis endpoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 476 | 520
score on a scale | 0.93 [0.00 to 6.00] | 1.06 [0.00 to 4.95]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.027, Wilcoxon Rank Sum Test; Median Difference (Final Values) = -0.13, 95% CI [-0.2 to 0.0]

5. Secondary Outcome: Average Rhinoconjunctivitis DMS Over the Entire GPS
Description: For rhinoconjunctivitis DMS, participants reported their use of specific rescue medications with specific scores assigned to each medication (score range: 0 to 36), with a lower score representing less use of medications for rhinoconjunctivitis.
Time Frame: Entire GPS (expected average duration of 5 to 6 weeks)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 629 | 672
score on a scale | 0.88 (0.11) | 1.36 (0.16)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.0003, Zero-Inflated Log-Normal Model — A zero-inflated log-normal mixed distribution model was used with treatment, baseline asthma status, age category (<18 or >=18 years) and pollen region as covariates; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.73 to -0.22]

6. Secondary Outcome: Average Rhinoconjunctivitis DSS Over the Peak GPS
Description: as for outcome 2
Time Frame: Peak GPS (expected average duration of 2 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 620 | 663
score on a scale | 2.71 [0.00 to 18.00] | 3.40 [0.00 to 17.57]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Median Difference (Final Values) = -0.69, 95% CI 2-sided [-0.9 to -0.2]

7. Secondary Outcome: Average Rhinoconjunctivitis DMS Over the Peak GPS
Description: as for outcome 5
Time Frame: Peak GPS (expected average duration of 2 weeks)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 620 | 663
score on a scale | 1.01 (0.13) | 1.63 (0.19)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.0001, Zero-Inflated Log-Normal Model — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.94 to -0.31]

8. Secondary Outcome: Average Paediatric Standardised Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Overall Score Over the Peak GPS (Participants 6 to <12 Years of Age)
Description: For PRQLQ, participants assessed a total of 19 items within 5 domains: Nose Symptoms, Eye Symptoms, Practical Problems, Activity Limitation and Other Symptoms, each on a scale of 0 to 6 (0=Not troubled, 6=Extremely troubled; score range: 0 to 6 [mean of all domain scores]), with a higher score indicating more significant impairment due to seasonal allergic rhinoconjunctivitis.
Time Frame: Peak GPS (expected average duration of 2 weeks)
Population: The FAS population consisted of all randomized participants <12 years of age who received at least one dose of study drug and had at least one post-treatment observation for the analysis endpoint.entry.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 13 | 12
score on a scale | 0.89 [0.00 to 2.36] | 0.75 [0.22 to 2.98]
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.644, Wilcoxon Rank Sum Test; Median Difference (Final Values) = 0.15, 95% CI 2-sided [-0.4 to 0.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 30 days after last dose of study drug (up to a total of 31 weeks).
Description: The Safety Population consisted of all randomized participants who received at least one dose of study treatment. Three randomized participants never received study drug and two participants were randomized to receive Placebo but actually received SCH 697243 instead.
Arm/Group | SCH 697243 | Placebo
Serious Adverse Events (participants affected / at risk) | 14/753 | 9/745
Other Adverse Events (participants affected / at risk) | 480/753 | 316/745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=753) | Placebo (N=745)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=753) | Placebo (N=745)
Ear pruritus (Ear and labyrinth disorders) | 92 (108) | 12 (13)
Lip swelling (Gastrointestinal disorders) | 46 (61) | 5 (5)
Oedema mouth (Gastrointestinal disorders) | 98 (126) | 9 (10)
Oral pruritus (Gastrointestinal disorders) | 139 (171) | 21 (24)
Paraesthesia oral (Gastrointestinal disorders) | 92 (152) | 24 (28)
Tongue pruritus (Gastrointestinal disorders) | 53 (66) | 5 (5)
Nasopharyngitis (Infections and infestations) | 103 (133) | 122 (148)
Upper respiratory tract infection (Infections and infestations) | 78 (97) | 86 (99)
Headache (Nervous system disorders) | 65 (100) | 56 (94)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (73) | 43 (49)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 39 (41) | 25 (28)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 (53) | 27 (37)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 181 (250) | 29 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the SPONSOR 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.